CLINICAL TRIAL: NCT05929807
Title: A Phase 2, Multicenter, Long-Term, Open Label Extension Trial Evaluating Safety, Tolerability, and Efficacy of Subcutaneous Doses of TransCon CNP Administered Once Weekly in Children and Adolescents With Achondroplasia
Brief Title: A Clinical Trial to Investigate Long-term Safety, Tolerability, and Efficacy of Weekly Subcutaneous Doses With TransCon CNP in Children and Adolescents With Achondroplasia
Acronym: AttaCH
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ascendis Pharma Growth Disorders A/S (Industry)
Responsible Party: Sponsor
Organization: Ascendis Pharma A/S (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASND0039
Record Dates: First submitted 2023-06-06; First posted 2023-07-03 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Achondroplasia
Keywords: Achondroplasia; Dwarfism
MeSH Terms: conditions — Achondroplasia; Dwarfism

STUDY DESIGN:
Intervention Model Description: Patients will roll over from previous TransCON CNP clinical trials
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TransCon CNP 100 mcg (Experimental): TransCon CNP 100 mcg delivered once weekly by subcutaneous injection
  Interventions: Drug: TransCon CNP

INTERVENTIONS:
Drug: TransCon CNP — TransCon CNP drug product is a lyophilized powder in a single-use vial. Prior to use, the lyophilized powder is reconstituted with sterile water for injection and administered by subcutaneous injection via syringe and needle.

SUMMARY:
TransCon CNP administered once-weekly in children and adolescents with achondroplasia who have completed a prior TransCon CNP clinical trial. Participants who complete a prior TransCon CNP trial and meet all eligibility criteria will be invited to continue into the long-term open label extension trial to receive 100 µg CNP/kg/week of TransCon CNP. Trial treatment will be completed when the participant reaches 16 years of age for females and 18 years of age for males and have femur and tibial epiphyseal closure. TransCon CNP treatment will continue if femur and tibial epiphyseal closure is not confirmed at the age of 16 years for females, and 18 years for males. Treatment with TransCon CNP will be completed once femur and tibial epiphyseal closure is confirmed by radiographic imaging. The trial duration is individual for each trial participant. Visits will occur every 12-14 weeks throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Written, signed informed consent of the parent(s) or legal guardian(s) of the participant, and as required by the institutional review board/human research ethics committee/independent ethics committee (IRB/HREC/IEC). For participants who are below the age of consent, a written assent will be obtained in accordance with applicable requirements as required by IRB/HREC/IEC. Upon reaching the legal age of consent, depending on applicable requirements, these participants will be asked to give their own written consent.
* Participants with achondroplasia who have completed a clinical trial with TransCon CNP.
* Parent(s)/legal guardian(s) willing and able to administer weekly SC injections of TransCon CNP and to follow the protocol.
* Considered eligible based on the safety evaluations performed for evaluating stopping/holding rule criteria during the prior TransCon CNP clinical trial.

Exclusion Criteria:

* Known or suspected hypersensitivity to the investigational product or related products (trehalose, tris[hydroxymethyl]aminomethane, succinate, and methoxy polyethylene glycol [mPEG]).
* Have received any dose of prescription medications, investigational medicinal product (other than TransCon CNP).
* Sexually active female participants and female partners of male participants of childbearing potential not using a highly effective form of contraceptive (including oral, injectable, or implantable contraception, or intrauterine device (IUD)) for the entire trial period and for 90 days post end of the trial.
* Participants with serum 25-hydroxy-vitamin D (25OHD) levels of <50 nmol/L (<20 ng/mL) at Visit 1 must be on treatment regimen of Vitamin D supplementation.
* Any disease or condition that, in the opinion of the investigator, may make the participant unlikely to fully complete the trial, may confound interpretation of trial results, or may present undue risk from receiving trial treatment. This could include family situations, complications or manifestations, or medications that might impact safety or be considered confounding.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2039-01 (Estimated); Study Completion 2039-03 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | Through trial completion, an average of 10 years
  Incidence of Treatment-Emergent Adverse Events
Height Z-scores | Through trial completion, an average of 10 years
  Number of standard deviations

SECONDARY OUTCOMES:
Annualized Growth Velocity | Through trial completion, an average of 10 years
  cm per year

CONTACTS AND LOCATIONS:
Overall Officials: Claus Strange, Study Director — Ascendis Pharma A/S
Locations (17):
- United States (8):
  - Ascendis Pharma Investigational Site, Little Rock, Arkansas
  - Ascendis Investigational Site, Aurora, Colorado
  - Ascendis Investigational Site, Wilmington, Delaware
  - Ascendis Investigational Site, Saint Paul, Minnesota
  - Ascendis Pharma Investigational Site, Columbia Falls, Montana
  - Ascendis Pharma Investigational Site, Buffalo, New York
  - Ascendis Investigational Site, Houston, Texas
  - Ascendis Pharma Investigational Site, Madison, Wisconsin
- Ascendis Pharma Investigational Site, Parkville, Victoria, Australia
- Ascendis Investigational Site, Linz, Austria
- Ascendis Investigational Site, Montreal, Canada
- Ascendis Pharma Investigational Site, Copenhagen, Denmark
- Ascendis Investigational Site, Berlin, Germany
- Ascendis Pharma Investigational Site, Dublin, Ireland
- Ascendis Investigational Site, Auckland, New Zealand
- Ascendis Investigational Site, Coimbra, Portugal
- Ascendis Investigational Site, Vitoria-Gasteiz, Spain

IPD SHARING:
Plan to Share IPD: No